CLINICAL TRIAL: NCT06112145
Title: Are Rehabilitation Results in Flexor Tendon Zone II Injuries as Bad as Feared?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Nazife Kapan, Principal investigatör, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AŞH-MK-ÇS
Record Dates: First submitted 2023-10-27; First posted 2023-11-01 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Flexor Tendon Rupture; Hand Injuries; Rehabilitation
MeSH Terms: conditions — Hand Injuries | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group I (Experimental): Flexor tendon zon II rupture patients
  Interventions: Other: rehabilitation program
- group II (Experimental): Flexor tendon other zon rupture patients
  Interventions: Other: rehabilitation program

INTERVENTIONS:
Other: rehabilitation program — All fingers of the injured hand are fitted with a dorsal blocking orthosis. Early passive mobilization exercises in the form of passive flexion and extension and edema massage will be taught and it will be recommended to be applied every two hours during the day.

SUMMARY:
The hand is the basic functional organ of the human body and is responsible for complex tasks such as grasping and catching. It also plays an important role in a person's daily life, self-care activities and business life. When the flexor tendon system, which is necessary for the effective use of the hand, is damaged, it can cause physical, socioeconomic deterioration, mood disorders and permanent disabilities in the individual. Treatment of flexor tendon injuries after appropriate surgical repair ıt includes an intensive rehabilitation program. In this study, it was aimed to investigate the early rehabilitation results of patients who underwent a rehabilitation program after Zone II flexor tendon injury by comparing the improvements in joint range of motion, pain, functionality and quality of life with other zone injuries.

DETAILED DESCRIPTION:
Tendon cuts constitute a significant portion of hand injuries. Today, most flexor tendon ruptures are repaired the same day as the injury or a few days later. Rehabilitation after flexor tendon repair is at least as important as surgical repair. Hand rehabilitation protocol after tendon repair; It consists of four periods: 1-4 weeks early period, 4-6 weeks early intermediate period, 6-8 weeks intermediate period, 8-12 weeks late period. Modified Duran Protocol is one of the earliest passive mobilization methods. According to this protocol, it has been reported that 3-5 mm of passive movement of the tendon anastomosis is effective in preventing tendon adhesions. In the literature, the number of studies examining rehabilitation results in patients with flexor tendon zone II injuries is quite limited. Post-operative rehabilitation results are worse in patients with zone II tendon injuries compared to other flexor zone injuries. This study aimed to investigate the early rehabilitation results of patients who underwent a rehabilitation program after Zone II flexor tendon injury by comparing the improvements in joint range of motion, pain, functionality and quality of life with other zone injuries. 70 patients who applied to Ankara City Hospital Physical Therapy and Rehabilitation Hospital Traumatic Hand Clinic due to flexor tendon injury and met the inclusion criteria for the study will be included. Demographic characteristics of the patients (age, gender), occupation, cause of injury, injured hand, dominant hand, smoking, and injury zones will be recorded. Patients with zone II injuries Group I, Patients with other zone injuries will be divided into Group II. In this study, Modified Duran early passive mobilization protocol was used to protect the repaired tendon and reduce the risk of adhesion will be followed. The physiotherapist will advised each patient on the things to consider after the operation, orthosis use and care, and the rehabilitation process. Early passive mobilization exercises in the form of passive flexion and extension and edema massage will be taught to all fingers of the injured hand in a dorsal blocking orthosis and will be recommended to be applied every two hours during the day. Patient follow-up will last four weeks and afterwards, measurements will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Had a traumatic flexor tendon injury
* In the acute period after repair (1-4 weeks)

Exclusion Criteria:

* Accompanying fracture, dislocation, burn
* infection, malignancy
* Patients using steroid-nonsteroidal drugs and having cognitive dysfunction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | baseline and 4th week
  Pain intensity of patients at rest and during activity will be evaluated with a visual analog scale (VAS). For VAS evaluation, the meanings of the numbers from 0 to 10 placed on a 10 cm line were explained to the patients. It will be announced that no pain is 0 points, moderate pain is 5 points, and the most severe pain is 10 points. According to these explanations, the patient will be asked to mark the pain on a 10 cm line. Pain intensity will be determined by measuring the distance between the marked place and the starting point with a ruler.
Range of motion | baseline and 4th week
  Range of motion is one of the most commonly used outcome variables after hand tendon injuries and will be preferred because it provides objective information about the effectiveness of the treatment. Since this study covers the acute period after repair, the normal joint movement of the patients will be evaluated passively. The measurement will be made with a goniometer.

SECONDARY OUTCOMES:
Duruoz Hand Index | baseline and 4th week
  Duruoz Hand Index is a self-reported measure of the patient's self-reported hand movements in the kitchen, while dressing, performing personal hygiene, at work, and other general movements. It consists of 18 items on skills. Scores range from 0 to 40 for kitchen work, from 0 to 10 for dressing, hygiene and office work, and from 0 to 20 for the "other" category. Patients rated their abilities as 0 (no difficulty) and 5 (impossible) to reach a total score between 0-90. A higher score represents greater activity restriction and more difficulty.
Short Form-36 | baseline and 4th week
  It is a 36-question scale consisting of physical function, physical role difficulty, emotional role difficulty, pain, vitality, general health and mental health subscales. Each subscale; It is scored so that "0" indicates the lowest and "100" indicates the best level of quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Nazife K KAPAN, MD, Principal Investigator — Kırşehir Ahi Evran University, Kırşehir/TURKEY; Merve K KAPAN, PT, Principal Investigator — Ankara City Hospital, Ankara/TURKEY; Berat Meryem A ALKAN, Prof. Dr., Study Director — Ankara City Hospital, Ankara/TURKEY; Bedriye B BAŞKAN, Prof. Dr., Study Director — Ankara City Hospital, Ankara/TURKEY; Tezel YŞ YILDIRIM ŞAHAN, Assoc. Prof., Study Director — Health Sciences Univercity, Gülhane faculty of physiotherapy and rehabilitation, Ankara/TURKEY
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Stenekes MW, Geertzen JH, Nicolai JP, De Jong BM, Mulder T. Effects of motor imagery on hand function during immobilization after flexor tendon repair. Arch Phys Med Rehabil. 2009 Apr;90(4):553-9. doi: 10.1016/j.apmr.2008.10.029. PMID 19345768
- [Background] Kannas S, Jeardeau TA, Bishop AT. Rehabilitation following zone II flexor tendon repairs. Tech Hand Up Extrem Surg. 2015 Mar;19(1):2-10. doi: 10.1097/BTH.0000000000000076. PMID 25700105
- [Background] Tang JB. Indications, methods, postoperative motion and outcome evaluation of primary flexor tendon repairs in Zone 2. J Hand Surg Eur Vol. 2007 Apr;32(2):118-29. doi: 10.1016/J.JHSB.2006.12.009. Epub 2007 Feb 12. PMID 17298858
- [Background] Cetin A, Dincer F, Kecik A, Cetin M. Rehabilitation of flexor tendon injuries by use of a combined regimen of modified Kleinert and modified Duran techniques. Am J Phys Med Rehabil. 2001 Oct;80(10):721-8. doi: 10.1097/00002060-200110000-00003. PMID 11562553